CLINICAL TRIAL: NCT01853384
Title: A Phase 3 Randomized Safety and Efficacy Trial of HP802-247 in the Treatment of Chronic Venous Leg Ulcers (EU)
Brief Title: Safety and Efficacy Trial of HP802-247 in the Treatment of Chronic Venous Leg Ulcers
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: based on outcome of trial NCT01656889.
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 802-247-09-032; 2012-003286-18 (EudraCT Number)
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Results first posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Venous Ulcer; Venous Stasis Ulcer; Ulcer
Keywords: Venous leg ulcer; ulcer; venous stasis; compression; venous; venous stasis ulcer; vlu; wound; varicose veins; venous insufficiency; dvt; deep vein thrombosis
MeSH Terms: conditions — Varicose Ulcer; Ulcer; Wounds and Injuries; Varicose Veins; Venous Insufficiency; Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HP802-247 plus compression therapy (Experimental): HP802-247 (fibrinogen solution & thrombin solution containing living, irradiated, growth arrested keratinocytes and fibroblasts) 260 µL (130 µL, one spray, of each solution) containing 0.5 X 10(6th) cells per mL every 14 days. Subjects randomized to HP802-247 will receive Vehicle on alternate weeks.
  Interventions: Biological: HP802-247
- HP802-247 Vehicle plus compression therapy (Placebo Comparator): fibrinogen solution & thrombin solution without cells. Subjects randomized to HP802-247 Vehicle will receive Vehicle weekly.
  Interventions: Other: HP802-247 Vehicle

INTERVENTIONS:
Biological: HP802-247 — Study Dosage / Usage: 260 µL (130 µL, one spray, of each solution) containing 0.5 X 10(6th) cells per mL every 14 days.
  Arms: HP802-247 plus compression therapy
Other: HP802-247 Vehicle — HP802-247 Vehicle consists of two separate components, a fibrinogen solution (Component 1) and a cell free thrombin solution which is identical to Component 2 except that no keratinocytes and no fibroblasts are present. A single dose is created when combined on the wound surface.
  Other Names: Placebo
  Arms: HP802-247 Vehicle plus compression therapy

SUMMARY:
This study is being done to find out if an investigational product called HP802-247 can help people with venous leg ulcers. Investigational means that HP802-247 has not been approved by the U.S. Food and Drug Administration (FDA).

This research is being done to compare the efficacy of HP802-247 plus compression therapy against Vehicle plus compression therapy in achieving complete wound closure over the 12-week treatment period. Vehicle looks the same as HP802-247 but contains no cells.

At least 440 subjects will participate. The study is going to be conducted in approximately 5 countries at approximately 50 sites across the European Union.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent.
* Age ≥ 18 years and of either sex.
* Willing to comply with protocol instructions, including allowing all study assessments.
* Have a venous leg ulcer (VLU) between the knee and ankle (at or above the malleolus), with a surface area ≥ 2.0 cm2 and ≤ 12.0 cm2
* Venous insufficiency confirmed by duplex Doppler ultrasound examination for valvular or venous incompetence.
* Arterial supply adequacy confirmed
* Target ulcer involves a full thickness skin loss, but WITHOUT exposure of tendon, muscle, or bone.
* Target ulcer duration ≥ 6 weeks but ≤ 104 weeks (24 months).
* Acceptable state of health and nutrition

Exclusion Criteria:

* History of anaphylaxis, serum sickness, or erythema multiforme reaction to aprotinin, bovine serum albumin or bovine serum proteins, penicillin, streptomycin, amphotericin B.
* Prior diagnosis of Systemic Lupus Erythematosus with elevated anti-DNA antibody titers, Buerger's disease (thromboangiitis obliterans), current diagnosis of vasculitis, or current diagnosis of claudication.
* Therapy with another investigational agent within thirty (30) days of Screening, or during the study.
* A target ulcer of non-venous etiologies (e.g., sickle cell anemia, necrobiosis lipoidica diabeticorum, pyoderma gangrenosum, vasculopathic or vasculitic).
* Documented history of osteomyelitis at the target wound location within 6 months preceding the Screening Visit.
* Refusal of or inability to tolerate compression therapy.
* Therapy of the target ulcer with autologous skin graft, Apligraf™, or Dermagraft™ within 30 days preceding the Screening Visit.
* History of cancer in the preceding 5 years (other than carcinoma in situ of the cervix or adequately treated non-melanoma skin cancers).
* Any prior exposure to HP802-247 or its vehicle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B. Slade, MD, Study Chair — Smith & Nephew, Inc.; Tommy Lee, MSHS, Study Director — Smith & Nephew, Inc.; Wolfgang Vanscheidt, Professor Dr, Principal Investigator — University Freiburg-Practice for Dermatology
Locations (46):
- Belgium (5):
  - Anderlecht
  - Brussels
  - Edegen
  - Ghent
  - Kortrijk
- Czechia (9):
  - Brno
  - Hradec Králové
  - Olomouc
  - Pardubice
  - Plzen-Bory
  - Prague
  - Třebíč
  - Uherské Hradiště
  - Ústí nad Labem
- Germany (15):
  - Bochum
  - Bonn
  - Cologne
  - Dresden
  - Düsseldorf
  - Essen
  - Freiburg im Breisgau
  - Göttingen
  - Greifswald
  - Hamburg
  - Kiel
  - Krefeld
  - Magdeburg
  - München
  - Münster
- Hungary (7):
  - Budapest
  - Debrecen
  - Hatvan
  - Orosháza
  - Sátoraljaújhely
  - Szeged
  - Szolnok
- Poland (10):
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Rzeszów
  - Studzionka
  - Warsaw
  - Wroclaw
  - Zabrze

REFERENCES:
- [Derived] Marston WA, Ennis WJ, Lantis JC 2nd, Kirsner RS, Galiano RD, Vanscheidt W, Eming SA, Malka M, Cargill DI, Dickerson JE Jr, Slade HB; HP802-247 Study Group. Baseline factors affecting closure of venous leg ulcers. J Vasc Surg Venous Lymphat Disord. 2017 Nov;5(6):829-835.e1. doi: 10.1016/j.jvsv.2017.06.017. PMID 29037354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 47 sites in the EU [Belgium (3), Czech Republic (8), Germany (15), Hungary (8), Poland (13)] between January 10, 2014 and November 27, 2014; sites included independent and hospital wound clinics and private practice sites.
Pre-assignment Details: Subjects entered a 2-week run-in; subjects whose wound radius decreased by < 0.349 cm/2weeks and met all other inclusion/exclusion (I/E) criteria were eligible for randomization. After completion of the treatment period, subjects entered a three-month follow up period.
Groups:
- HP802-247 Plus Compression Therapy: HP802-247 (fibrinogen solution & thrombin solution containing living, irradiated, growth arrested keratinocytes and fibroblasts) 260 µL (130 µL, one spray, of each solution) containing 0.5 X 10(6th) cells per mL every 14 days for up to 12 weeks or wound closure, which ever occurred first. Subjects randomized to HP802-247 will receive Vehicle on alternate weeks.
  HP802-247: Study Dosage / Usage: 260 µL (130 µL, one spray, of each solution) containing 0.5 X 10(6th) cells per mL every 14 days.
- HP802-247 Vehicle Plus Compression Therapy: fibrinogen solution & thrombin solution without cells. Subjects randomized to HP802-247 Vehicle will receive Vehicle weekly for up to 12 weeks or wound closure, which ever occurred first.
  HP802-247 Vehicle: HP802-247 Vehicle consists of two separate components, a fibrinogen solution (Component 1) and a cell free thrombin solution which is identical to Component 2 except that no keratinocytes and no fibroblasts are present. A single dose is created when combined on the wound surface.
Period: Randomized
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Started | 131 | 121
Completed | 69 | 75
Not Completed | 62 | 46
Not completed — Adverse Event | 5 | 3
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Sponsor Decision | 47 | 34
Not completed — Other | 3 | 3
Period: Enrolled in Follow up Period
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Started | 96 | 94
Not Enrolled in Follow-up | 35 | 27
Completed | 96 | 94
Not Completed | 0 | 0
Period: Completed Follow up Visit 1
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Started | 96 | 94
Completed | 82 | 85
Not Completed | 14 | 9
Not completed — Early Termination | 13 | 9
Not completed — Withdrawal by Subject | 1 | 0
Period: Completed Follow up Visit 2
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Started | 96 | 94
Completed | 93 | 91
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy | Total
Number analyzed (Participants) | 131 | 121 | 252
Age, Continuous [Mean (Full Range); unit: years] | 65.6 [28 to 90] | 68.1 [28 to 92] | 66.8 [28 to 92]
Age, Customized [Number; unit: participants]
  18-39 years | 6 | 3 | 9
  40-49 years | 6 | 3 | 9
  50-59 years | 26 | 20 | 46
  60-69 years | 40 | 40 | 80
  70+ years | 53 | 55 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 63 | 139
  Male | 55 | 58 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 129 | 120 | 249
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 131 | 121 | 252
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Compare the Treatment Groups for the Number of Subjects With Complete Wound Closure Over the 12-Week Treatment Period From Baseline
Description: For each treatment group the area of each subject's target ulcer was measured on a weekly basis, for up to 12 weeks, using a laser-based wound imaging system in conjunction with software to measure area. Following initial closure subjects returned for four weekly visits to confirm wound closure. Wounds that remained closed for four weeks were classified as confirmed closures; if a wound opened at any of the 4 visits it was not considered to have closed.
  For subjects who dropped from the study prior to the end of treatment, their remaining visit values were imputed using LOCF; wound status of closed was not imputed.
Time Frame: Weekly, over 12 Weeks or until wound closure, which ever occurred first
Population: ITT Populations: Subjects who received at least one dose of test article.
Measure: Number; unit: participants
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Number analyzed (Participants) | 131 | 121
participants
  Wounds Closed | 61 | 61
  Wounds Not Closed | 70 | 60
Statistical Analysis 1: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = .5348, Cochran-Mantel-Haenszel — Analysis adjusted for sites, with significance being at P < 0.05

2. Secondary Outcome: Compare the Efficacy of the Treatment Groups in Achieving Complete Wound Closure, Based on Time in Days to Closure Over the 12-Week Treatment Period From Baseline.
Description: This key secondary outcome was based on a Cox Proportional Hazard Analysis.
Time Frame: 12 Weeks
Population: ITT Populations: Subjects who received at least one dose of test article. Data were analyzed using the Cox Proportional hazard procedure, with significance being at P < 0.05.
Measure: Median (Full Range); unit: days
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Number analyzed (Participants) | 131 | 121
days | 57.0 [8.0 to 115.0] | 50.0 [6.0 to 134.0]
Statistical Analysis 1: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = .9456, Regression, Cox

3. Secondary Outcome: Compare the Efficacy of the Treatment Groups in Achieving Complete Wound Closure, Based on Median Time (Days) to Closure Over the 12-Week Treatment Period From Baseline.
Description: This key secondary outcome was based on a Kaplan-Meier Survival analysis.
Time Frame: 12 weeks
Population: ITT Populations: Subjects who received at least one dose of test article. Data were analyzed using Kaplan-Meier Survival analysis, with significance being at P < 0.05.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Number analyzed (Participants) | 131 | 121
days | 64 [57 to 78] | 57 [50 to 71]

4. Secondary Outcome: Compare the Treatment Groups for the Proportion of Subjects With Wound Closure at Each of the 12-Week Treatment Period From Baseline
Description: For subjects who dropped from the study, their remaining visit values were imputed using LOCF. Treatment groups were compared for percentage of participants with closed wounds at each treatment visit.
Time Frame: Weekly, over the 12 week treatment period, or until wound closure, which ever occurred first
Population: ITT Populations: Subjects who received at least one dose of test article. Analysis was by the Cochrane Mantel Haenszel (CMH) test, adjusted for sites, with significance being at P < 0.05
Measure: Number; unit: percentage of participants
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Number analyzed (Participants) | 131 | 121
percentage of participants
  Baseline | 0 | 0
  Treatment Week 01 | 2.3 | 3.3
  Treatment Week 02 | 8.4 | 7.4
  Treatment Week 03 | 13.7 | 18.2
  Treatment Week 04 | 22.1 | 25.6
  Treatment Week 05 | 26.7 | 33.9
  Treatment Week 06 | 29.8 | 38.0
  Treatment Week 07 | 32.8 | 39.7
  Treatment Week 08 | 37.4 | 39.7
  Treatment Week 09 | 38.9 | 43.8
  Treatment Week 10 | 40.5 | 46.3
  Treatment Week 11 | 41.2 | 47.9
  Treatment Week 12 | 48.1 | 53.7
  Week 12 - Primary Endpoint | 46.6 | 50.4
Statistical Analysis 1: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = .6194, Cochran-Mantel-Haenszel — Treatment Week 01
Statistical Analysis 2: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = .7930, Cochran-Mantel-Haenszel — Treatment Week 02
Statistical Analysis 3: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.3362, Cochran-Mantel-Haenszel — Treatment Week 03
Statistical Analysis 4: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.5263, Cochran-Mantel-Haenszel — Treatment Week 04
Statistical Analysis 5: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.1997, Cochran-Mantel-Haenszel — Treatment Week 05
Statistical Analysis 6: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.1617, Cochran-Mantel-Haenszel — Treatment Week 06
Statistical Analysis 7: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.2611, Cochran-Mantel-Haenszel — Treatment Week 07
Statistical Analysis 8: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.7232, Cochran-Mantel-Haenszel — Treatment Week 08
Statistical Analysis 9: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.4405, Cochran-Mantel-Haenszel — Treatment Week 09
Statistical Analysis 10: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.3516, Cochran-Mantel-Haenszel — Treatment Week 10
Statistical Analysis 11: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.2821, Cochran-Mantel-Haenszel — Treatment Week 11
Statistical Analysis 12: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.3722, Cochran-Mantel-Haenszel — Treatment Week 12
Statistical Analysis 13: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.5348, Cochran-Mantel-Haenszel — Week 12 - Primary Endpoint

5. Secondary Outcome: Number of Subjects With Durable Wound Healing Over the 3 Months Following Complete Wound Closure
Description: Subjects who completed the treatment period with confirmed wound closure were followed in the post-treatment period for a further two months to determine their closed wound status (remained closed/reopened), giving a measure of persistence of wound closure following completion of treatment.
Time Frame: Target ulcer status observed at two (visit 1) and three (visit 2) months following initial ulcer closure.
Population: Due to study termination the data available to assess durability of closure were limited to only the subjects who completed at least one of the follow-up visits. Participants who had CLOSED wounds at completion of treatment; 103 subjects (HP802-247: 49; Vehicle: 54) completed Visit 18, 114 subjects (HP802-247: 57; Vehicle: 57) completed Visit 19
Measure: Number; unit: participants
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Number analyzed (Participants) | 134 | 132
participants
  Follow-up Visit 1 (wounds remained closed) | 45 | 52
  Follow-up Visit 1 (wounds reopened) | 4 | 2
  Follow-up Visit 2 (wounds remained closed) | 51 | 47
  Follow-up Visit 2 (wounds reopened) | 6 | 10

6. Secondary Outcome: Change From Baseline in Pain Associated With the Target Wound at Each of the 12 Double Blind Treatment Weeks
Description: Target ulcer pain was measured using a Visual Analog Scale [Range: 0mm - 100mm]. Subjects marked their pain level on a 100 mm horizontal line, with a short vertical line across the scale, 0 denoting no pain and 100mm the maximum pain.
Time Frame: Baseline and Weekly, over the 12 week treatment period
Population: ITT Populations: Subjects who received at least one dose of test article. Data were analyzed by an ANCOVA, adjusted for site and baseline score.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Number analyzed (Participants) | 131 | 121
mm
  Baseline | 29.40 (28.5) | 26.30 (28.3)
  Week 01 | -8.6 (2) | -7.5 (2.1)
  Week 02 | -10.4 (2.2) | -11.0 (2.3)
  Week 03 | -14.0 (2.3) | -10.7 (2.4)
  Week 04 | -14.3 (2.3) | -12.1 (2.3)
  Week 05 | -17.2 (2.1) | -13.6 (2.2)
  Week 06 | -17.8 (2.2) | -15.4 (2.2)
  Week 07 | -18.5 (2.0) | -17.5 (2.1)
  Week 08 | -20.0 (2.0) | -17.1 (2.1)
  Week 09 | -19.7 (2.1) | -17.9 (2.1)
  Week 10 | -18.9 (2.0) | -18.4 (2.1)
  Week 11 | -19.4 (2.0) | -19.7 (2.1)
  Week 12 | -20.0 (2.0) | -20.1 (2.0)
Statistical Analysis 1: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.5909, ANCOVA — Week 01
Statistical Analysis 2: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.8234, ANCOVA — Week 02
Statistical Analysis 3: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.1556, ANCOVA — Week 03
Statistical Analysis 4: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.3487, ANCOVA — Week 04
Statistical Analysis 5: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.1064, ANCOVA — Week 05
Statistical Analysis 6: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.2888, ANCOVA — Week 06
Statistical Analysis 7: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.6095, ANCOVA — Week 07
Statistical Analysis 8: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.1566, ANCOVA — Week 08
Statistical Analysis 9: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.4216, ANCOVA — Week 09
Statistical Analysis 10: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.8166, ANCOVA — Week10
Statistical Analysis 11: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.9114, ANCOVA — Week 11
Statistical Analysis 12: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.9733, ANCOVA — Week 12

7. Secondary Outcome: Change From Baseline in Pain Associated With the Target Leg at Each of the 12 Double Blind Treatment Weeks
Description: Target leg pain were measured using a Visual Analog Scale [Range: 0mm - 100mm]. Subjects marked their pain level on a 100 mm horizontal line, with a short vertical line across the scale, 0 denoting no pain and 100mm the maximum pain.
Time Frame: Baseline and Weekly, over the 12 week treatment period
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Number analyzed (Participants) | 131 | 121
mm
  Baseline | 24.18 (27.0) | 22.35 (16.0)
  Week 01 | -4.1 (2.3) | -4.9 (2.4)
  Week 02 | -2.2 (2.3) | -1.3 (2.4)
  Week 03 | -9.2 (2.2) | -5.3 (2.3)
  Week 04 | -10.1 (2.2) | -8.8 (2.2)
  Week 05 | -9.7 (2.3) | -8.6 (2.3)
  Week 06 | -12.2 (2.0) | -9.1 (2.1)
  Week 07 | -13.1 (2.2) | -8.9 (2.2)
  Week 08 | -14.2 (2.1) | -9.0 (2.1)
  Week 09 | -10.1 (2.2) | -6.3 (2.3)
  Week 10 | -12.7 (2.1) | -11.1 (2.2)
  Week 11 | -12.9 (2.0) | -11.8 (2.1)
  Week 12 | -14.3 (2.0) | -12.2 (2.1)
Statistical Analysis 1: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.7439, ANCOVA — Week 01
Statistical Analysis 2: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.6992, ANCOVA — Week 02
Statistical Analysis 3: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.0867, ANCOVA — Week 03
Statistical Analysis 4: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.5739, ANCOVA — Week 04
Statistical Analysis 5: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.6497, ANCOVA — Week 05
Statistical Analysis 6: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.1427, ANCOVA — Week 06
Statistical Analysis 7: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.0682, ANCOVA — Week 07
Statistical Analysis 8: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.0161, ANCOVA — Week 08
Statistical Analysis 9: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.0973, ANCOVA — Week 09
Statistical Analysis 10: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.4661, ANCOVA — Week 10
Statistical Analysis 11: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.6010, ANCOVA — Week 11
Statistical Analysis 12: Comparison: HP802-247 Plus Compression Therapy vs HP802-247 Vehicle Plus Compression Therapy; Test type: Superiority or Other; p = 0.3369, ANCOVA — Week 12

ADVERSE EVENTS:
Time Frame: Up to 19 Weeks or subjects who completed 12 weeks of treatment and the post-treatment follow up. For subjects who had wound closure, collection time included the treatment period and the post-treatment period
Description: All subjects randomized to treatment were questioned about adverse events and were included in the number of participants assessed for safety. The first assessments at each weekly visit were about changes in general health and concomitant medications and the occurrence of adverse events.
Arm/Group | HP802-247 Plus Compression Therapy | HP802-247 Vehicle Plus Compression Therapy
Serious Adverse Events (participants affected / at risk) | 5/131 | 12/121
Other Adverse Events (participants affected / at risk) | 60/131 | 64/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP802-247 Plus Compression Therapy (N=131) | HP802-247 Vehicle Plus Compression Therapy (N=121)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (2)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Wound sepsis (Infections and infestations) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HP802-247 Plus Compression Therapy (N=131) | HP802-247 Vehicle Plus Compression Therapy (N=121)
Gastrointestinal disorders (Gastrointestinal disorders) | 5 (9) | 6 (8)
General disorders and administration site conditions (General disorders) | 3 (3) | 9 (11)
Infections and infestations (Infections and infestations) | 15 (20) | 19 (23)
Infected skin ulcer (Infections and infestations) | 7 (9) | 5 (7)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 18 (22) | 13 (13)
Excoriation (Injury, poisoning and procedural complications) | 10 (12) | 6 (6)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 9 (13) | 14 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 12 (15)
Nervous system disorders (Nervous system disorders) | 2 (7) | 4 (4)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 30 (62) | 39 (87)
Dermatitis (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (6)
Skin maceration (Skin and subcutaneous tissue disorders) | 2 (3) | 7 (13)
Skin ulcer (Skin and subcutaneous tissue disorders) | 17 (34) | 20 (37)
Venous ulcer pain (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Vascular disorders (Vascular disorders) | 5 (8) | 10 (11)
Hypertension (Vascular disorders) | 5 (8) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less